CLINICAL TRIAL: NCT01005680
Title: A Randomized Phase 3 Study Comparing Pemetrexed Plus Cisplatin With Gemcitabine Plus Cisplatin as First-Line Treatment in Patients With Advanced Non-squamous Non-Small Cell Lung Cancer.
Brief Title: A Study Comparing Two Different Chemotherapy Types in Chinese Patients With Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12878; H3E-CR-JMIL (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed plus Cisplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin
- Gemcitabine plus Cisplatin (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 milligrams/square meter (mg/m²) administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
  Other Names: Alimta; LY231514
  Arms: Pemetrexed plus Cisplatin
Drug: Gemcitabine — 1250 mg/m² administered intravenously on Day 1 and Day 8 of each 21-day cycle, for 6 cycles
  Other Names: Gemzar; LY188011
  Arms: Gemcitabine plus Cisplatin
Drug: Cisplatin — 75 mg/m² administered intravenously on day 1 of each 21 day cycle, for 6 cycles

SUMMARY:
The purpose of this study is to compare the efficacy and safety of two different chemotherapy types in the first line treatment of advanced Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Present with histologically proven or cytological diagnosis of non-squamous non-small cell lung cancer (NSCLC) Stage IIIB or IV.
* Participants must agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug.
* Female participants must not be pregnant.
* No prior systemic chemotherapy for lung cancer.
* At least one unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Adequate organ function.
* Prior radiation therapy allowed to <25% of the bone marrow.
* Signed informed consent document on file.
* Estimated life expectancy of greater than or equal to 12 weeks.
* Participant compliance and geographic proximity that allow adequate follow up.

Exclusion Criteria:

* Peripheral neuropathy of great than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the participant's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Documented brain metastases unless the participant has completed successful local therapy for central nervous system metastases and has not taken corticosteroids for at least 4 weeks before enrollment.
* Presence of clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.
* Significant weight loss (that is, greater than or equal to 10%) over the previous 6 weeks before study entry.
* Concurrent administration of any other anti-tumor therapy.
* Inability to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Inability to take corticosteroids.
* Pregnant or breast-feeding.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- China (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dalian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sichuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed Plus Cisplatin (PC): Pemetrexed: 500 milligrams/square meter (mg/m²) administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
  Cisplatin: 75 mg/m² administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
- Gemcitabine Plus Cisplatin (GC): Gemcitabine: 1250 mg/m² administered intravenously on Day 1 and Day 8 of each 21-day cycle, for 6 cycles
  Cisplatin: 75 mg/m² administered intravenously on Day 1 of each 21-day cycle, for 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Started | 126 | 130
Received at Least 1 Dose of Study Drug | 125 | 127
Completed | 120 | 119
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Gemcitabine Plus Cisplatin (GC): Gemcitabine: 1250 mg/m² administered intravenously on Day 1 and day 8 of each 21-day cycle, for 6 cycles
  Cisplatin: 75 mg/m² administered intravenously on day 1 of each 21 day cycle, for 6 cycles
- Total: Total of all reporting groups
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC) | Total
Number analyzed (Participants) | 126 | 130 | 256
Age Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.65) | 55.7 (9.95) | 56.1 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 59 | 114
  Male | 71 | 71 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 126 | 130 | 256
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 126 | 130 | 256
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 126 | 130 | 256

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from date of randomization to date of death from any cause. Participants who were alive were censored at the date of last contact.
Time Frame: Randomization to date of death from any cause up to 35.8 months post-randomization
Population: Intent-to-Treat: all participants and are analyzed according to the treatment group they were randomly assigned. Censored participants: PC=37, GC=39.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 126 | 130
months | 17.54 [13.34 to 22.67] | 15.51 [13.70 to 19.29]
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.822, Cox Proportional Hazard — HR adjusted for treatment, disease stage, Eastern Cooperative Oncology Group Performance Status (ECOG PS), sex, and basis for initial pathological diagnosis; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.77 to 1.39]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the date of randomization to date of first observation of clinical or objective progressive disease (PD) or death due to any cause. PD assessed using Response Evaluation Criteria in Solid Tumor (RECIST v1.0) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of one or more new lesions. Participants who were not known to have died or had PD were censored at the date of last contact.
Time Frame: Randomization to first date of Progressive Disease (PD) or death from any cause up to 33.0 months post-randomization
Population: Intent-to-Treat: all randomized participants who are analyzed according to the treatment group they were randomly assigned. Censored participants: PC=8, GC=10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 126 | 130
months | 5.88 [4.99 to 6.47] | 5.85 [5.59 to 6.41]
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.640, Cox Proportional Hazard — HR adjusted for treatment, disease stage, Eastern Cooperative Oncology Group Performance Status (ECOG PS), sex and basis for initial pathological diagnosis; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.82 to 1.37]

3. Secondary Outcome: Time to Progressive Disease (TtPD)
Description: TtPD defined as the time from study randomization to the first date of progressive disease (PD). PD assessed using Response Evaluation Criteria in Solid Tumor (RECIST v1.0) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of 1 or more new lesions. Participants who were not known to have PD or who died without PD were censored at the date of last of last tumor assessment.
Time Frame: Randomization to first date of PD up to 23.7 months post-randomization
Population: Intent-to-Treat: all randomized participants who were analyzed according to the treatment group they were randomly assigned. Censored participants: PC=12, GC=19.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 126 | 130
months | 5.82 [4.76 to 6.47] | 5.82 [5.55 to 6.34]
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.928, Cox Proportional Hazard — HR adjusted for treatment, disease stage, Eastern Cooperative Oncology Group Performance Status (ECOG PS), sex and biases for initial pathological diagnosis; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.78 to 1.32]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from first objective status assessment of complete response (CR) or partial response (PR) to the first time progressive disease (PD) or death as a result of any cause. Response using Response Evaluation Criteria in Solid Tumor (RECIST v1.0) criteria. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Participants who are not known to have died or to have PD were censored at the date of last contact. PD assessed using RECIST v1.0 and defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of 1 or more new lesions
Time Frame: Date of first response to the date of (PD) or death from any cause up to 22.9 months post-randomization
Population: Intent-to-Treat: all randomized participants who were analyzed according to the treatment group they were randomly assigned and who achieved CR or PR. Censored participants: PC=1, GC=0.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 30 | 24
months | 4.53 [4.17 to 5.88] | 4.98 [3.55 to 6.41]
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.887, Cox Proportional Hazard — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.51 to 1.79]

5. Secondary Outcome: Time to Treatment Failure (TtTF)
Description: TtTF was defined as date of randomization until the date of discontinuation of study treatment due to adverse event, progressive disease (PD), or death from any cause. PD assessed using Response Evaluation Criteria in Solid Tumor (RECIST v1.0) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of 1 or more new lesions. Participants who discontinued study treatment for any other reason were censored at the date of discontinuation of study treatment. Participants still on study drug at data-inclusion cut-off date were censored at the cut-off date.
Time Frame: Randomization until date of discontinuation of study treatment due to adverse events, PD, or death from any cause up to 6.3 months post-randomization
Population: Intent-to-Treat: all randomized participants who were analyzed according to the treatment group they were randomly assigned. Censored participants: PC=85, GC=91.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 126 | 130
months | NA [NA to NA] — Results were not calculable due to high censoring rate. | NA [NA to NA] — Results were not calculable due to high censoring rate.
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.861, Cox Proportional Hazard — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.67 to 1.61]

6. Secondary Outcome: Tumor Response Rate
Description: Tumor response rate was the percentage of participants with confirmed best tumor response of complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumor (RECIST v1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions; Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions. Progressive disease (PD) assessed using RECIST v1.0 criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of 1 or more new lesions.
Time Frame: Randomization until date of objective PD or death from any cause up to 35.8 months post-randomization
Population: Tumor Response-Qualified Population: all randomized participants who received at least l dose of study drug, who were diagnosed with locally advanced/metastatic non-small cell lung cancer, who had at least 1 baseline and 1 post-baseline tumor measurement, and who were not on concurrent systemic chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 121 | 116
percentage of participants | 24.8 | 20.7
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.451, two-sided Z test

7. Secondary Outcome: Risk/Benefit Ratio
Description: Risk/benefit ratio was calculated as the percentage of participants who experienced a study-drug related toxicity of Common Terminology Criteria for Adverse Events (CTCAE v3.0) Cancer Therapy Evaluation Program (CTEP) Grade 3 or higher, divided by the Kaplan-Meier estimated percentage of participants surviving one year.
Time Frame: Randomization to date of death from any cause up to 35.8 months post-randomization
Population: Safety population: all randomized participants who received at least 1 dose of study drug and were analyzed according to actual treatment received in Cycle 1 of 21-day cycle.
Measure: Number; unit: ratio
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 125 | 127
ratio | 0.70 | 0.83

8. Other Pre Specified Outcome: Disease Control Rate (DCR)
Description: DCR was the percentage of participants with Complete Response (CR), Partial Response (PR), and Stable Disease (SD). Response determined using Response Evaluation Criteria In Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target lesions; PR was defined as at least a 30% decrease in sum of longest diameter of target lesions; progressive disease (PD) was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter ever recorded since study treatment started, or the appearance of 1 or more new lesions; SD was defined as small changes that did not meet the above criteria.
Time Frame: Randomization to date of objective PD or death from any cause up to 35.8 months post-randomization
Population: Tumor Response Qualified Population: all randomized participants who received at least l dose of study drug, who were diagnosed with locally advanced/metastatic non-small cell lung cancer, who had at least 1 baseline and 1 post-baseline tumor measurement, and who are not on concurrent systemic chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 121 | 116
percentage of participants | 78.5 | 75.9
Statistical Analysis 1: Comparison: Pemetrexed Plus Cisplatin (PC) vs Gemcitabine Plus Cisplatin (GC); Test type: Superiority or Other; p = 0.627, two-sided Z test

9. Other Pre Specified Outcome: Survival Without Toxicity (SWT)
Description: SWT was defined as the time from randomization to a study-drug related toxicity. Toxicity was defined as Common Terminology Criteria for Adverse Events (CTCAE v3.0) Grade 3 or 4 or death. Participants who do not have a CTCAE Grade 3 or higher toxicity and are alive will be censored at the date of last contact.
Time Frame: Randomization to date of toxicity or date of death up to 34.6 months post-randomization
Population: Safety population: all randomized participants who received at least 1 dose of study drug and were analyzed according to actual treatment received in Cycle 1 of 21-day cycles. Censored participants: PC=22, GC=10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Number analyzed (Participants) | 125 | 127
months | 5.85 [4.21 to 8.38] | 2.56 [1.68 to 3.78]

ADVERSE EVENTS:
Arm/Group | Pemetrexed Plus Cisplatin (PC) | Gemcitabine Plus Cisplatin (GC)
Serious Adverse Events (participants affected / at risk) | 8/125 | 9/127
Other Adverse Events (participants affected / at risk) | 120/125 | 123/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Cisplatin (PC) (N=125) | Gemcitabine Plus Cisplatin (GC) (N=127)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Cisplatin (PC) (N=125) | Gemcitabine Plus Cisplatin (GC) (N=127)
Anaemia (Blood and lymphatic system disorders) | 28 (32) | 44 (54)
Leukopenia (Blood and lymphatic system disorders) | 53 (101) | 60 (142)
Lymphopenia (Blood and lymphatic system disorders) | 8 (11) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 52 (122) | 65 (148)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (18) | 13 (23)
Constipation (Gastrointestinal disorders) | 21 (29) | 32 (47)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 8 (10)
Dyspepsia (Gastrointestinal disorders) | 6 (9) | 8 (12)
Nausea (Gastrointestinal disorders) | 56 (132) | 59 (131)
Vomiting (Gastrointestinal disorders) | 44 (95) | 54 (88)
Fatigue (General disorders) | 33 (66) | 33 (55)
Pyrexia (General disorders) | 10 (10) | 9 (10)
Alanine aminotransferase increased (Investigations) | 25 (36) | 24 (32)
Aspartate aminotransferase increased (Investigations) | 20 (27) | 13 (20)
Blood creatinine increased (Investigations) | 5 (6) | 7 (9)
Blood sodium decreased (Investigations) | 10 (16) | 11 (14)
Haemoglobin decreased (Investigations) | 21 (24) | 33 (47)
Neutrophil count decreased (Investigations) | 28 (69) | 30 (68)
Platelet count decreased (Investigations) | 4 (4) | 16 (28)
Red blood cell count decreased (Investigations) | 5 (8) | 7 (8)
White blood cell count decreased (Investigations) | 25 (59) | 32 (68)
Decreased appetite (Metabolism and nutrition disorders) | 46 (88) | 39 (67)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (14) | 10 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (21) | 7 (11)
Dizziness (Nervous system disorders) | 8 (13) | 5 (7)
Insomnia (Psychiatric disorders) | 7 (7) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 15 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days